CLINICAL TRIAL: NCT03830697
Title: The Trial Was Completed by Shaanxi Provincial Hospital of Traditional Chinese Medicine and Northwest Women and Children's Hospital. Thirty-five Patients With POR Who Underwent ART (Assisted Reproductive) Treatment Were Observed in Each Center. Patients in the Experimental Group Were Given Acupuncture Treatment for 12 Weeks Prior to COH. If the Patient Has a Good COH Timing During Acupuncture Treatment, She Will Enter the COH Cycle at Any Time. Patients in the Control Group Waiting for 12 Weeks Before COH
Brief Title: A Trial Study on Acupuncture Treatment of Poor Ovarian Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaanxi Hospital of Traditional Chinese Medicine (Other)
Collaborators: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-11-29
Record Dates: First submitted 2018-12-19; First posted 2019-02-05 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-11

CONDITIONS: Poor Ovarian Response

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menstruation situation TCM symptom score standard (Experimental)
  Interventions: Other: Acupuncture intervention
- Sham intervention (Placebo Comparator)
  Interventions: Other: Acupuncture intervention

INTERVENTIONS:
Other: Acupuncture intervention — Patients in the experimental group were given acupuncture treatment for 12 weeks prior to COH. If the patient has a good COH timing during acupuncture treatment, he or she will enter the COH cycle at any time.The acupuncture intervention program of the test group is as follows:Acupoint group 1: Baihui（DU20）, Zhongyu（RN12）, Tianshu （ST25）(bilateral), Guanyuan（RN4）, uterus (bilateral)（EX-CA1）, Dahe（KI12） (bilateral),Zusanli （ST36）(bilateral), Sanyinjiao（SP6） (bilateral), Taichong （LR3）(both sides).

SUMMARY:
The trial was completed by Shaanxi Provincial Hospital of Traditional Chinese Medicine and Northwest Women and Children's Hospital. Thirty-five patients with POR who underwent ART (Assisted Reproductive) treatment were observed in each center. Patients in the experimental group were given acupuncture treatment for 12 weeks prior to COH. If the patient has a good COH timing during acupuncture treatment, she will enter the COH cycle at any time. Patients in the control group waited for 12 weeks before COH. In this study, the COH regimen of the two groups of patients was the same, and the appropriate ovulation induction protocol was selected by the investigator according to the B-ultrasound and endocrine conditions of the patient's menstrual day 1-3. At the end of treatment, patients were observed for the number of eggs in the COH cycle, fertilization rate, cleavage rate, available embryo rate, high quality embryo rate, implantation rate, ovarian reserve function assessment, menstrual status and peri-menopausal symptoms.

DETAILED DESCRIPTION:
1.Acupuncture intervention

1. test group Patients in the experimental group were given acupuncture treatment for 12 weeks prior to COH. If the patient has a good COH timing during acupuncture treatment, he or she will enter the COH cycle at any time.

   The acupuncture intervention program of the test group is as follows:

   Acupoint group 1: Baihui（DU20）, Zhongwan（RN12）, Tianshu （ST25）(bilateral), Guanyuan（RN4）, uterus (bilateral)（EX-CA1）, Dahe（KI12） (bilateral),Zusanli （ST36）(bilateral), Sanyinjiao（SP6） (bilateral), Taichong （LR3）(both sides) Acupoint group 2： Baihui（DU20）,ShenShu（BL23）、ZhongLiao（BL33）、TaiXi（KI3） Operation: The two-point group was used alternately, with the group 1 as the initial treatment. The patient took the appropriate position (point group 1 was taken in the supine position, group 2 was taken in the prone position), and the local skin of the acupoint was routinely disinfected. Baihui, flat thorn 0.5-1.0 inch; Tai Chong, acupuncture 0.5-1.0 inch in the direction of Yongquan; Shenshu, Taixi, straight thorn 0.5-1.0 inch; ZhongLiao（BL33） , inward and downward oblique thorn 2.0-2.5 inch, It is required to puncture the hole in the second hole; the remaining hole is straight 1.0-1.5 inch. All the acupoints are evenly inserted and twisted (the Baihui acupoints only turn around). Each time the needle is kept for 20 minutes, once every other day, 3 times a week for a total of 12 weeks.
2. Control group Patients in the control group waited for 12 weeks before COH。

2.Standard IVF/ICSI Process

1. COH process（In this study, the COH regimen was the same in both groups, and the investigator chose the antagonist regimen based on the B-ultrasound and endocrine conditions on the 1-3 day of menstruation.） 1）Gn start time: Menstruation Day3 days, B-ultrasound and hormone levels (FSH/LH/E2/P/β-HCG) suggest that the ovary is in a basal state; 2）Gn starting dose: 75~300 IU; 3）Gn dose adjustment: 5 days after administration, according to ovarian response (B-ultrasound and E2 levels) Whole Gn dose, hMG (Hemeiqi) can be added if necessary; 1 ovarian response is monitored every 1~2 days thereafter (B-ultrasound and E2 level), adjust the amount of Gn accordingly。 4）When the antagonist is added: when the dominant follicle is ≥12mm, add antagonist (Eugly) 250ug/d to HCG day (including HCG day); 5）HCG trigger timing and dose: at least 3 follicles ≥ 18mm, given HCG4000~8000IUim.
2. Eggs taken 36 hours after intramuscular injection of HCG:
3. In vitro fertilization, embryo culture:In vitro fertilization was performed 4 to 6 hours after egg retrieval, and Day 3 embryos were scored according to the general standards of each center.The two embryos with the highest score were labeled as the embryos of the first embryo transfer. The remaining embryos are often Freeze on Day3, Day5 or Day6.
4. Embryo transfer and corpus luteum support：On Day 3, the patient maintained bladder filling and transplanted 2 of the best quality under the guidance of transabdominal B-ultrasound.Embryo; or on day 5, under the guidance of transabdominal B-ultrasound, transplant 1-2 blastocysts; continue to gestrinone 20mg Bid po supports the corpus luteum.
5. Pregnancy test： 1）Determination of blood βHCG levels 14 days after ET or Cryopreserved embryo transfer (CET) to determine biochemical pregnancy; 2）If determined to be pregnant, continue corpus luteum support。 3）35 days after ET, determine the clinical pregnancy by transvaginal B-ultrasound, record the number of gestational sacs, location, large Small, the presence or absence of fetal buds, the presence or absence of fetal heart, other abnormal conditions.

ELIGIBILITY:
Inclusion Criteria:

1. POR compliant diagnostic criteria
2. Intracytoplasmic sperm injection, ICSI）。 Indication with IVF or intracytoplasmic sperm injection (ICSI).

3.18≤age<40

Exclusion Criteria:

1. Repeated spontaneous abortion 2 or more patients (including biochemical pregnancy abortion.
2. Patients who have failed to undergo repeated implantation (at least 3 transplanted transplants, at least 3-6 high-quality embryos without clinical pregnancy);
3. uterine malformation (single uterus, double uterus, double uterus, untreated mediastinal uterus) and other effects affecting uterine cavity disease (adenomyosis, submucosal uterine fibroids, intrauterine adhesions and scar uterus) Patient;
4. Patients and their husbands with abnormal karyotypes (excluding chromosomal polymorphisms;
5. Untreated patients with hydrosalpinx;
6. (6)Patients with contraindications to ART and pregnancy, or those with a clear influence on pregnancy, such as hypertension, clinically symptomatic heart disease, diabetes, liver disease, kidney disease, severe anemia, history of venous thrombosis, History of pulmonary embolism or cerebrovascular events, history of malignant tumors;
7. Refusal to sign the informed consent form.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of eggs obtained in the COH cycle. | After an average of 13 days in the COH cycle
  The number of eggs obtained in the controlled ovarian hyperstimulation cycle.

SECONDARY OUTCOMES:
Ovarian reserve function assessment | 12 week
  Basal sinus follicle count AFC, AMH and basal hormone levels (package)Including FSH, LH and E2)
Chinese Medicine Symptoms Scoring Standard for Menstruation | 12 week
  Menstrual situation:Mainly assess the menstrual cycle and menstrual flow. menstrual cycle is based on the results of the patient's own comparison.Divided into normal cycle, early menstruation (>7 days before menstruation) and delayed menstruation (>7 days after menstruation) 3class. According to the patient's own comparison results, the menstrual volume is divided into normal menstruation and less menstrual flow.Reduce, or the menstrual period is less than 2 days, or even a drop. It is generally believed that the amount of menstruation is less than 20ml for less menstruation.Class 2.
Self-RatingAnxietyScale | 12 week
  Menstrual disorders, less menstrual flow, hot flashes, night sweats or cold, convulsions, forgetfulness, irritability Insomnia, secondary symptoms include dizziness, tinnitus, dull complexion, waist and knee pain, itchy skin, low libido.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi, China